CLINICAL TRIAL: NCT01440036
Title: The Correlation Between the Enzyme Paraoxigenase 1 (PON1) to Carotid Artery Atheromatous Plaque
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, yehudit.hackmon, Principal Investigator, Ziv Hospital
Other Study IDs: 0032-11-ZIV
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery; Atherosclerotic plaque; paraoxygenase 1 PON1; Patients undergoing carotid artery endarterectomy CEA for carotid artery stenosis
MeSH Terms: conditions — Carotid Stenosis; Plaque, Atherosclerotic | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Atherosclerotic plaque from carotid arteries Blood sample (5cc)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid endarterectomy: Patients that have the common indication for the treatment of carotid artery stenosis by surgery - CEA (carotid endarterectomy), symptomatic and asymptomatic patients.
  Interventions: Procedure: Carotid endarterectomy

INTERVENTIONS:
Procedure: Carotid endarterectomy — The removal of atherosclerotic plaque from the carotid artery, by surgery

SUMMARY:
The objective of the research, is to examine the hypothesis, that the enzyme paraoxygenase 1 ( PON1) can influence carotid artery's atherosclerotic plaque content and stability, and its relation to plasma's enzyme concentration.

DETAILED DESCRIPTION:
Atherosclerosis is a major risk factor for morbidity and mortality in the western world. It is characterized by the accumulation of fat (cholesterol) in the arterial wall, creation of the atheromatous plagues and the creation of arterial stenosis and occlusion. The cellular content of theses plaques include: fibroblasts, endothelial cells, smooth muscle cells, macrophages, and lipids: phospholipids, cholesterol, oxysterols and fatty acids. Lipids penetration from the blood stream collaborates different proteins, including the anti-atherogenic enzyme - paraoxygenase 1 - PON1. This enzyme has many ani-atherogenic activities, e.g. Protection from oxygenation and increase of cholesterol efflux from macrophages by HDL. Although the enzyme has a verity of substrates and known anti-atherogenous function, its mechanism is still vogue. The enzymes accumulation rate is the function of the advancement of the fatty strike towards advanced lesion. There is evidence that the presence accumulation and activity of the PON1 within the plaque, is a defense mechanism against atherosclerosis development. The assumption to be proved is that PON1 can control plaque's content and influence its atherogenous factors. Furthermore, we will try to identify these factors that the PON1 acts on. Beside plaque's content and PON1's influence on them, we would like to investigate the phenotype of haptoglobin in the subjects that the plaques were removed from. It is known that diabetics that have the genotype haptoglobin 2-2, characterized by increased risk for oxygenation stress and cardiovascular events (up to 5 times). We would like to examine if there is a correlation between plaque's content, PON1's ability to disassemble oxygenized factors within the plaque, and the phenotype to haptoglobin.

Methods: The plaque source will be from carotid endarterectomy, in the vascular unit. This procedure is a routine operation for patients suffering from carotid artery stenosis, based on clinical decisions. The plaques will be transported to a lipid laboratory soon after they will be harvested, will be frozen in liquid nitrogen and processed into powder. This material will be the origin for the proteins we try to extract. Patient's blood samples (that is drawn routinely for the operation) will be the source for the characterization of the haptoglobin's genotype.

It is critical to emphasize that routinely, the plaques are waste products, and only 5 cc of additional blood is withdrawn from the patients for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CEA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CEA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2014-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel, Israel